CLINICAL TRIAL: NCT05955846
Title: A Prospective Multicenter Clinical Trial to Evaluate the Safety and Effectiveness of an Intraocular Lens With a Virtual Aperture Optic
Brief Title: Evaluation of Safety and Effectiveness of an IOL With a Virtual Aperture Optic
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Z Optics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VAO-IOL-004
Record Dates: First submitted 2023-07-03; First posted 2023-07-21 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Intraocular Lens; Cataract; Presbyopia
MeSH Terms: conditions — Cataract; Presbyopia | interventions — Cataract Extraction

STUDY DESIGN:
Intervention Model Description: Prospective, Single arm, Four centers study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Z+ VAO IOL (Experimental): FG-80030.1 hydrophobic
  Interventions: Procedure: cataract surgery; Device: implantation of device IOL FG-80030.1

INTERVENTIONS:
Procedure: cataract surgery — Subjects will undergo surgery to remove cataract (natural cloudy lens) via phacoemulsification implant the IOL Both eyes will be treated one month apart. Subjects will be followed up during 12 months
Device: implantation of device IOL FG-80030.1 — implant the IOL in both eyes. Both eyes will be treated one month apart. Subjects will be followed up during 12 months

SUMMARY:
Cataracts are cloudy areas in the lens of the eye that can cause changes in vision. Symptoms of cataracts include cloudy or fuzzy vision and sensitivity to glare. Cataract extraction with Intraocular lens (IOL) implantation is the most commonly performed surgical procedure in the world.

Presbyopia affects almost everyone over the age of 50. With age, the natural crystalline lens loses its ability to change shape, or accommodate, to focus on near distances. Thus, individuals with excellent distance vision will still need to wear spectacles for near tasks such as reading, and intermediate tasks such as computer work.

DETAILED DESCRIPTION:
The Z+ Virtual Aperture Optic IOL has been designed to perform similarly to monofocal IOL in that it corrects for distance vision but is also designed to provide a greater depth of focus. This greater depth of focus should improve near and intermediate visual acuities and thus reducing spectacle dependance. Therefore, it is expected that the Z+ Virtual Aperture Optic IOL will be a safe and efficient option for patients with presbyopia who desires spectacle independence after cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Adults, Age 40 to 75 years at the time of surgery, diagnosed with bilateral cataracts with planned cataract removal by phacoemulsification with a clear cornea incision and posterior chamber IOL implantation;
2. Preoperative best-corrected distance visual acuity (BCDVA) worse than 20/30 Snellen;
3. Clear intraocular media, other than cataract;
4. Calculated lens power within the available range (available range of +16 D to +24 D);
5. Preoperative keratometric astigmatism of less than 0.75 D in both operative eyes;
6. Potential for postoperative BCDVA of 20/25 or better in each eye after cataract removal and IOL implantation;
7. Able to comprehend and have signed a statement of informed consent;
8. Availability, willingness, ability and sufficient cognitive awareness to comply with examination procedures and study visits;

Exclusion Criteria:

1. Desire for monovision correction
2. History of Dry Eye treatments/devices (example IPL, Lipiflow, iLux, Tear Care, Bruder Mask, True Tear) or any dry eye medications other than artificial tears (example, Restasis, Xiidra, Cequa, Klarity-C, generic cyclosporine/compounded cyclosporine)
3. Active or recurrent anterior segment pathology (chronic uveitis, iritis, iridocyclitis, rubeosis iridis, Reiter's syndrome, etc.);
4. Clinically significant corneal abnormalities or defects including corneal dystrophy (e.g., epithelial, stromal, or endothelial dystrophy), irregularity (including irregularity due to dry eye syndrome), inflammation or edema per the Investigator's expert medical opinion. Note: conditions including, but not limited to: keratitis, keratoconjunctivitis, keratouveitis, keratopathy, or keratectasia should be excluded;
5. Previous corneal or intraocular surgery;
6. Irregular corneal astigmatism; or regular corneal astigmatism greater than or equal to +/-0.75D;
7. Inability to achieve stable keratometric readings for contact lens wearers;

   *The recommended time for discontinued wear of extended-wear or daily wear soft lenses is one week prior to surgery, one month for gas permeable and six months for PMMA lenses. No evidence of significant corneal warpage from contact lens use should be present on corneal topography and if the subject has been wearing a rigid gas permeable contact lens there should be two stable serial topographies at least 1 month following cessation of contact lens wear
8. Higher-order Zernike corneal aberrations (3rd -order and above) RMS value greater than 1.0 um for the central 6-mm diameter area;
9. Pupil dilation in scotopic conditions >5mm
10. Use of systemic or ocular medications that may affect vision or likely to impact pupil dilation or iris structure;
11. Pharmacologically dilated pupil size less than 6 mm in either eye;
12. Pupil abnormalities;
13. History of ocular trauma, prior refractive or other ocular surgery or subjects expected to require retinal laser treatment or other surgical intervention;
14. Any disease or pathology, other than cataract, that (in the expert opinion of the Investigator) is expected to reduce the potential postoperative BCDVA. Note: Conditions including, but not limited to the following: amblyopia, clinically severe corneal dystrophy (e.g., epithelial, stromal, or endothelial dystrophy), diabetic retinopathy, extremely shallow anterior chamber, not due to swollen cataract, microphthalmos, previous retinal detachment, previous corneal transplant, recurrent severe anterior or posterior segment inflammation of unknown etiology, iris; neovascularization, uncontrolled glaucoma, aniridia, or optic nerve atrophy, or diagnosis of pseudoexfoliation;
15. Neovascularization, uncontrolled glaucoma, aniridia, or optic nerve atrophy;
16. Subjects who have profound sensitivity to glare at night with oncoming traffic headlights or subjects who are sensitive to fluorescent light flicker;
17. Subjects who may reasonably be expected to require a SSI at any time during the study (other than YAG capsulotomy);
18. Subject is pregnant, plans to become pregnant, is lactating or has another condition associated with hormonal fluctuation that could lead to refractive changes and dry eye. Females of childbearing age must have a negative pregnancy test at screening in order to be enrolled into the study.
19. Concurrent participation or participation in any clinical trial up to 30 days prior to preoperative visit;
20. Acute, chronic, or uncontrolled systemic or ocular disease or any illness that, in the opinion of the investigator, would increase the operative risk or confound the outcome(s) of the study (e.g., poorly-controlled diabetes);

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Binocular photopic uncorrected visual acuity | 6 months
  * Binocular photopic uncorrected visual acuity at 6-months at 4 meters (infinity): uncorrected distance visual acuity (UDVA).
  * Binocular photopic uncorrected visual acuity at 6-months at 4 meters (infinity) at 66 cm (intermediate): uncorrected intermediate visual acuity (UIVA).
  * Binocular photopic uncorrected visual acuity at 6-months at 4 meters (infinity) at 1.5 meters (intermediate walking visual acuity): uncorrected walking visual acuity (UWVA)

SECONDARY OUTCOMES:
Efficacy : Binocular defocus/depth of focus curve | 3 months
  Binocular defocus/depth of focus curve under photopic conditions at the 3-month visit. Depth of Focus is calculated as the mean binocular diopters of range of focus where the visual acuity is 20/40 or better. The depth of focus will be measured at 66 cm, using the UIVA as the starting point. Defocus will be measured in 0.50D steps from +1.5D of positive defocus to -2.5D of negative defocus.
Efficacy : Uncorrected Visual Acuity | 6 months
  3 meters (TV viewing distance): uncorrected TV visual acuity (UTVVA) at 6 months.
Efficacy : Visual Acuity | 1 month
  * VA under mesopic conditions at 1.5m using ETDRS charts.
  * VA under mesopic conditions at 66cm using ETDRS charts.
Efficacy : Continuous-objective visual assessment by Vivior defocus curves | 12 Months
  Continuous-objective visual assessment: Measured with Vivior Visual Behavior monitor and assessed with the Vivior defocus curves to compare post-operative vs pre-operative visual requirements
Efficacy : Patient questionnaire | 12 Months
  Patient reported outcomes: Near Activity Visual Questionnaire (NAVQ)
  Questions related to the difficulty of the patient to perform tasks at near distance. Evaluation is rated on a scale from 0 to 3 defined as follows :
  0 : No difficulty
  1. : A little difficulty
  2. : Moderate difficulty
  3. : Extrement difficulty
Safety - Best corrected visual acuity | 1 month
  Loss of 10 letters or more of BCDVA when compared to Loss of 10 letters or more of BCDVA when compared to Preoperative or Postop Month 1.
Safety : Visual Acuity | 1 month
  * VA under mesopic conditions at 1.5 m.
  * VA under mesopic conditions at 66cm.
Safety : Percentage of patient with visual disturbances | 12 Months
  Assessment of visual disturbances at 6-month visit using either the Glare/Halo simulator and/or an objective assessment of Visual Disturbance
Safety : secondary surgical interventions | 12 Months
  The cumulative rate of secondary surgical interventions (SSIs) related to the optical properties of the IOL
Safety : Intraocular Pressure (IOP) | 12 Months
  Intraocular Pressure (IOP)
Safety : Slit Lamp Examination | 12 Months
  * Evaluation of Lens centration.
  * Evaluation of lens tilt.
  * Examination of capsule.
  * Examination of striae ratings.
Safety : slit lamp observations | 12 Months
  IOL Observations including Posterior Capsule Opacification
Safety : Rate of Posterior Capsulotomy | 12 Months
  Rate of Posterior Capsulotomy
Safety : Slit lamp Fundus Visualization | 12 Months
  Fundus Visualization